CLINICAL TRIAL: NCT04413838
Title: Study of the Efficiency and Security of NIVOLUMAB Therapy, Used in Immuno-stimulation, in Hospitalized Obese Individuals at Risk to Evolve Towards Severe Forms of COVID-19 Infection. Multicentric, Paralleled, Randomized, Controlled Trial
Brief Title: Efficiency and Security of NIVOLUMAB Therapy in Obese Individuals With COVID-19(COrona VIrus Disease) Infection
Acronym: NIVISCO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0478
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Obesity, COVID-19 Infection
Keywords: COVID-19; Obesity; Nivolumab; Immunotherapy; Anti-PD1
MeSH Terms: conditions — Obesity; COVID-19 | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIVOLUMAB on top of routine standard of care (Experimental): This correspond to COVID-19+ patients diagnosed upon biological testing (PCR Coronavirus SARS-CoV2), hospitalized, obese (BMI≥30kg/m²), with low lymphocyte counts, without high biological probability of macrophage activation syndrome (hemoglobin < 9.2 g/dl AND a blood platelets < 110000/mm3 AND aspartate aminotransferase (AST) > 30 U/l AND ferritin > 600 mg/l) and upon oxygen (either using mask or nasal cannula) but without criteria for ICU admission benefiting from a NIVOLUMAB treatment and routine standard of care for COVID-19 infection at the time of study inclusion
  Interventions: Drug: NIVOLUMAB
- Standard of care for COVID-19 infection (Other): This correspond to COVID-19+ patients diagnosed upon biological testing (PCR Coronavirus SARS-CoV2), hospitalized, obese (BMI≥30kg/m²), with low lymphocyte counts, without high biological probability of macrophage activation syndrome (hemoglobin < 9.2 g/dl AND a blood platelets < 110000/mm3 AND AST > 30 U/l AND ferritin > 600 mg/l) and upon oxygen (either using mask or nasal cannula) but without criteria for ICU admission benefiting from a routine standard of care for COVID-19 infection at the time of study inclusion
  Interventions: Other: Routine standard of care

INTERVENTIONS:
Drug: NIVOLUMAB — IV injection within 30 minutes of 24ml file (=240 mg) containing NIVOLUMAB BMS(Bristol-Myers Squibb) 10mg/ml (immune check point inhibitor targeting PD-1) on top of routine standard of care for COVID-19 infection
  Arms: NIVOLUMAB on top of routine standard of care
Other: Routine standard of care — No intervention is planned in this arm. Patients will follow routine standard of care for the COVID-19 treatment
  Arms: Standard of care for COVID-19 infection

SUMMARY:
Although SARS-CoV-2 (Severe Acute Respiratory Syndrome-associated coronavirus) due to COVID-19 evolves poorly towards ARDS (Acute Respiratory Distress Syndrome) and death, there is to date no validated drug available for severe forms of COVID-19. Patients with COVID-19 undergo a drastic decrease of T lymphocytes (LT) count, while the remaining ones display an "exhausted" phenotype, due to immunosuppressive pathway activation among which the Programed cell Death 1 (PD1) receptor pathways. LT exhaustion is responsible for host anergy towards viral infection and leads to increased risk of severe forms of COVID-19. Moreover, while the number of systemic LT PD1+ correlates with poor prognosis clinical stages of COVID-19 infection, healing from COVID-19 associates with LT PD1 expression normalization. Chinese epidemiologic data identified clinical risk factors of poor clinical evolution (i.e. ARDS or death), among which is found obesity, similarly to observation previously obtained during H1N1 infection (flu virus).

Obese persons display meta-inflammation and immune dysfunction, a condition similar to ageing, thus termed "Inflamm-aging", thus also used during obesity. Inflamm-aging, characterized by cytotoxic LT exhaustion and reduced NK cell (Natural Killer cell) cytotoxic function secondary to PD1 pathway activation, could contribute to the poor prognosis observed during cancer and infection in obese individuals. We hypothesize that the immunocompromised profile observed during obesity contribute to their vulnerability towards COVID-19.

In cancer or certain infection diseases, NIVOLUMAB, an anti-PD1 monoclonal antibody, restores exhausted LT immunity. We thus hypothesize that NIVOLUMAB-induced immunity normalization could (i) stimulate anti-viral response also during COVID-19 infection and (ii) prevent ARDS development, which has previously been associated with low LT count concomitant with increased inflammatory cytokine production.

This randomized controlled therapeutic trial, using an add-on strategy to usual standard of care, aims at demonstrating the efficacy and safety of NIVOLUMAB-induced cytotoxic LT normalization, to improve clinical outcomes in hospitalized COVID-19+ adult obese individuals with low LT, since they are at risk of poor prognosis. We postulate that NIVOLUMAB will increase the number of individuals able to stop oxygen therapy at D15

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years old
* COVID-19+ patients diagnosed upon biological testing (PCR Coronavirus SARS-CoV2)
* Hospitalized patients
* Obese individuals (BMI≥30kg/m²)
* Lymphocyte counts between 500 and 1500/mm3.
* Patients upon oxygen (either using mask or nasal cannula).
* Patients within their first 7 days after the beginning of symptoms.
* Women of childbearing potential: effective contraception for the duration of the study and 5 months after the administration of treatment.
* Patient who understands and accepts the need for a long term follow-up,
* Patients who agrees to be included in the study and who signs the informed consent form,
* Patients affiliated to a healthcare insurance plan.

Exclusion Criteria:

* CRITERIA LINKED TO THE DISEASE SEVERITY :

  * Patients hospitalized in ICU or constant care unit.
  * Patients with clinical symptoms requiring ICU admission (respiratory rate>30/min, oxygen requirement> 4Liters/min (using high concentration mask) to reach and maintain O2saturation>90%, qSOFA≥ 2(quick score of Sepsis-related Organ Failure Assessment), or associated multi-visceral failure.
  * Patients with high biological probability of macrophage activation syndrome (hemoglobin < 9.2 g/dl AND a blood platelets < 110000/mm3 AND AST > 30 U/l AND ferritin > 600 mg/l).

CRITERIA LINKED TO THE TREATMENT TOXICITY :

* Patients currently treated for cancer or with personal history of cancer within the last 3 years.
* Patients with Chronic Obstructive Pulmonary Disease (COPD) (GOLD 3 and 4 stages).
* Chronic respiratory insufficiency treated with oxygen.
* Patients aged above 70 years old.
* Active smoking.
* Personal history of thoracic radiotherapy.
* Patients with known sensibility to NIVOLUMAB or one of its component.
* Patients upon immunosuppressive dosage of corticoids.
* Patients upon immunosuppressive therapy or immunosuppressed patients.
* Patients already presenting severe autoimmune disease, for whom additional immunologic activation response would potentially precipitate lethal prognosis

GENERAL CRITERIA:

* Minor Patients
* Mentally unbalanced patients, under supervision or guardianship,
* Patient deprived of liberty,
* Patient who does not understand French/ is unable to give consent,
* Patient already included in a trial who may interfere with the study or in a period of exclusion following participation in a previous study.
* Pregnant (controlled by a pregnancy test) or lactating woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Patient's clinical state | 15 days after randomization
  Patient's clinical state will be evaluated by the proportion of patients able to be weaned of oxygen at D15 after randomization (randomization date is the day where the experimental treatment (i.e. NIVOLUMAB) is administered).

SECONDARY OUTCOMES:
Readmission | 7 days and 15 days after randomization
  Proportion of in-coming patients in ICU at D7 and D15 post-randomization
Mortality | 7 days and 15 days after randomization
  Proportion of death at D7 and D15 post-randomization
Oxygen flow needs | 7 days after randomization
  Proportion of patients weaned out of oxygen at D7 post-randomization
Requirement of oxygen | 7 days and 15 days after randomization
  Mean oxygen flow needed
Discharge from hospital | 7 days and 15 days after randomization
  Proportion of out-coming patients from hospitalization at D7 and D15 post-randomization
Adverse events | Within 15 days post-randomization and 90 days and 6 months after randomization
  Report of all adverse events linked or not to experimental treatment during the study
Presence of nasopharyngeal SARS-CoV-2 | On day 0 before randomization and 15 days after randomization
  Presence or not of nasopharyngeal SARS-CoV-2 determined by PCR response
nasopharyngeal SARS-CoV-2 viral charge | On day 0 before randomization and 15 days after randomization
  Presence or not of nasopharyngeal SARS-CoV-2 Quantified by PCR
Number of total Lymphocytes T | On day 0 before randomization and 15 days after randomization
  Number of total LT (using immuno-phenotyping) will explore the immune response
Number of CD3+ Lymphocytes T(lymphocyte subpopulation of CD3+ T cells) | On day 0 before randomization and 15 days after randomization
  Number of CD3+ LT (using immuno-phenotyping) will explore the immune response
Number of CD4+ Lymphocytes T(lymphocyte subpopulation of CD4+ T cells) | On day 0 before randomization and 15 days after randomization
  Number of total CD4+ LT (using immuno-phenotyping) will explore the immune response
Number of CD8+ Lymphocytes T(lymphocyte subpopulation of CD8+ T cells) | On day 0 before randomization and 15 days after randomization
  Evaluation of number of CD8+ LT (using immuno-phenotyping) will explore the immune response
Interleukin 6 (IL-6) | On day 0 before randomization and 15 days after randomization
  Systemic concentration measurement of IL-6 will explore the inflammatory response
Interleukin 10 (IL-10) | On day 0 before randomization and 15 days after randomization
  Systemic concentration measurement of IL-10 will explore the inflammatory response
Tumor Necrosis Factor alpha (TNFα ) | On day 0 before randomization and 15 days after randomization
  Systemic concentration measurement of TNFα will explore the inflammatory response
Interferon gamma (IFNγ) | On day 0 before randomization and 15 days after randomization
  Systemic concentration measurement of IFNγ will explore the inflammatory response
Type I Interferon (type I IFN) | On day 0 before randomization and 15 days after randomization
  Systemic concentration measurement of type I IFN will explore the inflammatory response
Tim3 expression | On day 0 before randomization and 15 days after randomization
  Evaluation of Tim3 expression on CD4+ and CD8+ lymphocytes will explore the fundamental research on obesity and COVID-19
PD1 expression | On day 0 before randomization and 15 days after randomization
  Evaluation of PD1 expression on CD4+ and CD8+ lymphocytes will explore the fundamental research on obesity and COVID-19
PD-L1 expression | On day 0 before randomization and 15 days after randomization
  Measurement of PD-L1 expression on monocytes will explore explore the fundamental research on obesity and COVID-19
Human Leukocyte Antigen - DR isotype gene expression (HLA-DR expression) | On day 0 before randomization and 15 days after randomization
  Measurement of HLA-DR expression on monocytes will explore explore the fundamental research on obesity and COVID-19
Production of IFNγ by lymphocytes T | On day 0 before randomization and 15 days after randomization
  The cytotoxic LT production of IFNγ will explore the fundamental research on obesity and COVID-19
Production of granzyme B by lymphocytesT | On day 0 before randomization and 15 days after randomization
  The cytotoxic LT production of granzyme B will explore the fundamental research on obesity and COVID-19
Lipopolysaccharides (LPS) | On day 0 before randomization and 15 days after randomization
  Measurement of LPS will explore the endotoxemia and perform fundamental research on obesity and COVID-19
LBP(LPS-Binding Protein) | On day 0 before randomization and 15 days after randomization
  Measurement of LBP (endotoxin transporter) will explore the endotoxemia and perform fundamental research on obesity and COVID-19
sCD14 | On day 0 before randomization and 15 days after randomization
  Measurement of sCD14 (endotoxin transporter) will explore the endotoxemia and perform fundamental research on obesity and COVID-19
High Density Lipoproteins | On day 0 before randomization and 15 days after randomization
  Measurement of High Density Lipoproteins proteomic will explore the lipoprotein metabolism and perform fundamental research on obesity and COVID-19
Apolipoprotein | On day 0 before randomization and 15 days after randomization
  Measurement of apolipoprotein proteomic will explore the lipoprotein metabolism and perform fundamental research on obesity and COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud Service Endocrinologie, Diabète et Nutrition, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No